CLINICAL TRIAL: NCT05990023
Title: Investigating the Effect of Computerized Vestibular Function Assessment and Interactive Training System, Combined With Cognitive/Motor Dual-task for the Elderly With Dizziness
Brief Title: The Effect of Computerized Vestibular Function Assessment and Training System Combined With Cognitive/Motor Dual-task
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N202212070
Record Dates: First submitted 2023-05-22; First posted 2023-08-14 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-05

CONDITIONS: Vestibular Function Disorder; Cognitive Decline; Dizziness; Vestibular Abnormality
Keywords: Vestibular function; Elderly cognition; Vestibular functional assessment; Vestibular vertigo
MeSH Terms: conditions — Vestibular Diseases; Cognitive Dysfunction; Dizziness; Vertigo

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional vestibule rehabilitation training (Active Comparator): The intervention for the control group primarily follows conventional rehabilitation methods but incorporates the computerized training system developed in this project.
  Interventions: Other: Traditional vestibule rehabilitation training
- Dual-task vestibule rehabilitation training (Experimental): The intervention for the experimental group is based on the intervention for the control group, with additional components based on the findings from the second year of the study. These dual-task exercises are integrated into the training using the computerized training system and provided to the experimental group.
  Interventions: Other: Dual-task vestibule rehabilitation training

INTERVENTIONS:
Other: Traditional vestibule rehabilitation training — * Standing, using a gaze tracking system on a force plate to track a continuously moving target, with alerts when body sway exceeds a certain threshold.
  * Standing, wearing an inertial sensor on the head and performing left-right or up-down head movements while maintaining gaze on a target, with a screen providing feedback on head movement speed.
  * Standing, controlling body weight distribution on the force plate to reach a target position, with a screen displaying the current center of gravity position.
  * Walking, synchronizing head movements with a rhythm or performing up-down head nods, with auditory cues indicating the desired head movement frequency.
  * During continuous head rotations, stepping in a regular sequence of forward, backward, left, and right movements.
  Arms: Traditional vestibule rehabilitation training
Other: Dual-task vestibule rehabilitation training — * Adding a dual task of digit countdown and recitation to clinical balance training exercises.
  * Incorporating a numerical calculation task into interactive screens during clinical balance training, with the participant's responses input by the researchers.
  * Introducing upper limb exercises, such as button pressing or arm swinging, during clinical balance training.
  * During continuous head rotations, following visual prompts on the display to perform forward, backward, left, and right displacements.
  Arms: Dual-task vestibule rehabilitation training

SUMMARY:
This study aims to investigate the effect of computerized vestibular function assessment and interactive training system, combined with cognitive/motor dual-task for the elderly with dizziness. The investigators will compare the movement abilities among older adults with different cognitive level, and further establish an assessment module that can evaluate participants' dual-task performance in both vestibular and cognitive tasks. Finally, leveraging the advantages of sensor detection technology and computerized feedback, an appropriate dual-task rehabilitation approach for vestibular function and cognition will be developed.

DETAILED DESCRIPTION:
Dizziness is one of the most common complaints among older adults and often a concern within healthcare systems. It leads to distressing sensations, reduced mobility, and decreased quality of life. Dizziness is also closely associated with falls, which are a major cause of comorbidities and mortality in older adults. During clinical rehabilitation training, it has been observed that some elderly patients with vestibular dizziness often experience difficulties with speech clarity, lack of attention, poor direction control, or easy forgetfulness of rehabilitation training content. Similar observations have been made by scholars who interacted with dizzy patients, noting difficulties in maintaining attention, deficits in attention and spatial memory, speech expression impairments, and impacts on spatial memory, fluency of speech, thinking abilities, calculation impairments, and other forms of numerical cognition. Clinical studies have already noted the association between vestibular dysfunction and cognitive impairment. However, there is limited research that can clarify the intricacies and complexities of this issue. Currently, there is scarce knowledge regarding the relationship between the vestibular system and specific cognitive aspects, as well as its correlation with balance deficits.

This study aims to investigate the effect of computerized vestibular function assessment and interactive training system, combined with cognitive/motor dual-task for the elderly with dizziness. Drawing from previous clinical rehabilitation experiences, a method for assessing vestibular function and balance performance will be designed to compare the movement differences among older adults with different cognitive performances. Subsequently, through scientific and objective motion capture analysis, a comprehensive assessment module will be established to evaluate the dual-task performance of participants in both vestibular and cognitive tasks. The performance differences attributed to cognition will be analyzed, and the correlation with vestibular function performance will be integrated to serve as a prescription reference for computer-assisted rehabilitation interventions. Finally, leveraging the advantages of sensor detection technology and computerized feedback, an appropriate dual-task rehabilitation approach for vestibular function and cognition will be developed. Methods: First year, the study will recruit 60 elderly people and integrate the use of inertial sensors and force plates with vestibular and balance tests to establish a vertigo assessment system for the elderly. In the second year, the subjects were divided into two groups: a control group of 25 healthy elderly people, and an experimental group of 25 elderly people who had experienced dizziness and falls in the past two years. Data were collected using a motion analysis system combined with a computerized assisted assessment. The main analysis is whether the experience of dizziness or fall affects the balance, vestibular and cognitive related activities. In the third year, 40 vestibular hypofunction patients will be randomized into either traditional or dual-task group. Both groups will receive 2~3 times per week for 4 weeks of computerized vestibular interventions with and without dual-task training protocols. Expected achievements: Combining safe stochastic dual-task training and computer-assisted rehabilitation interventions in this 3-year project, the mechanisms of cognition related to vestibular training will be elucidated. The optimal strategy for vestibular rehabilitation can thus be established.

ELIGIBILITY:
Inclusion Criteria:

* Year 1 (Study A):

  1. Could walk more than 30 meters with or without walking aids independently.
  2. Able to comprehend and communicate in Mandarin or Taiwanese.
  3. Sufficient corrected vision that allows independent outdoor mobility.
* Year 2 (Study B):

  1. Could walk more than 30 meters with or without walking aids independently.
  2. Able to comprehend and communicate in Mandarin or Taiwanese.
  3. Sufficient corrected vision that allows independent outdoor mobility.
  4. Healthy participants and those who have experienced dizziness or falls within the past two years.
* Year 3 (Study C):

  1. Could walk more than 30 meters with or without walking aids independently.
  2. Able to comprehend and communicate in Mandarin or Taiwanese.
  3. Sufficient corrected vision that allows independent outdoor mobility.
  4. Willing to engage in moderate-intensity exercise for 45 minutes per session.
  5. Participants who have experienced dizziness or falls within the past two years.

Exclusion Criteria:

* Year 1 (Study A):

  1. Severe central or peripheral nervous system disorders.
  2. Participants who are blind or deaf.
  3. Individuals who cannot communicate or understand instructions.
  4. Current fractures or significant joint injuries.
* Year 2 (Study B):

  1. Severe central or peripheral nervous system disorders.
  2. Participants who are blind or deaf.
  3. Individuals who cannot communicate or understand instructions.
  4. Current fractures or significant joint injuries.
* Year 3 (Study C):

  1. Severe central or peripheral nervous system disorders.
  2. Participants who are blind or deaf.
  3. Individuals who cannot communicate or understand instructions.
  4. Current fractures or significant joint injuries.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-05-14 (Estimated)

PRIMARY OUTCOMES:
Rotation of head, chest, and pelvis. | 3 year.
  Parameters from inertial sensors placed on the head, chest, and pelvis will be extracted. The parameters include rotational angles (degrees) of the head, chest, and waist.
Inclination of head, chest, and pelvis. | 3 year.
  Parameters from inertial sensors placed on the head, chest, and pelvis will be extracted. The parameters include angular velocities (degrees per second) of the head, chest, and waist.
Acceleration of head, chest, and pelvis. | 3 year.
  Parameters from inertial sensors placed on the head, chest, and pelvis will be extracted. The parameters include accelerations (meters per second squared) of the head, chest, and waist.
Static Visual acuity. | 3 year.
  Parameters recorded by a screen with optotype chart and eyeglass system.
Dynamic Visual acuity. | 3 year.
  Parameters recorded by a screen with optotype chart and eyeglass system during movements.
Static vestibulo-ocular reflex (VOR gain) | 3 year.
  The VOR gain calculated by dividing eye movement velocity by head rotation velocity. The eye movement velocity(degree per second) and head rotation velocity(degree per second) are recorded by a screen, eyeglass system, and inertial sensor on subject's head.
Dynamic vestibulo-ocular reflex. (VOR gain) | 3 year.
  The VOR gain calculated by dividing eye movement velocity by head rotation velocity. The eye movement velocity(degree per second) and head rotation velocity(degree per second) are recorded by a screen, eyeglass system, and inertial sensor on subject's head during movements.
Step length (centimeter) during walking | 3 year.
  Step length (centimeter) recorded by wearable sensors (inertial movement unit) or optical motion sensors (camera) during flat ground walking and up/down stairs situation from the starting location.
Step frequency | 3 year.
  Steps and times recorded by wearable sensors (inertial movement unit) or optical motion sensors (camera) during flat ground walking and up/down stairs situation from the starting location.
Walking trajectory (centimeter) | 3 year.
  The shift(centimeter) of light and motion markers on subjects recorded by wearable sensors (inertial movement unit) or optical motion sensors (camera) during flat ground walking and up/down stairs situation from the starting location.
Step width (centimeter) during walking | 3 year.
  The medial-lateral distance(centimeter) of light and motion markers on subject's feet recorded by wearable sensors (inertial movement unit) or optical motion sensors (camera) during flat ground walking and up/down stairs situation among the testing session.
Step variability of step length (standard deviation) during walking | 3 year.
  The standard deviation of step length(centimeter) among the testing session. The step length(centimeter) is recorded by wearable sensors (inertial movement unit) or optical motion sensors (camera) during flat ground walking and up/down stairs situation.
Step variability of step width (standard deviation) during walking | 3 year.
  The standard deviation of step width(centimeter) among the testing session. The step width(centimeter) is recorded by wearable sensors (inertial movement unit) or optical motion sensors (camera) during flat ground walking and up/down stairs situation.
Speed (meter per second) during walking | 3 year.
  Speed (meter per second) calculated by dividing walking distances by total walking times. The walking distances and times are recorded by wearable sensors (inertial movement unit) or optical motion sensors (camera) during flat ground walking and up/down stairs situation from the starting location.
Lower limb Joint force (Newton) | 3 year.
  Joint force is calculated by joint position(millimeter) and ground reaction force(Newton). The joint position(millimeter) is recorded by wearable sensors (inertial movement unit) or optical motion sensors (camera), and ground reaction force(Newton) is recorded by forceplates.
Lower limb Joint moment (Newton-metre) | 3 year.
  Joint moment (Newton-metre) is calculated by multiplying ground reaction force(Newton) by limb length(meter). The limb length(meter) is recorded by meters or optical motion sensors(camera).
Lower limb Joint power (Watt) | 3 year.
  Joint Power(watt) is calculated as the "scalar product" of joint moment and joint angular velocity(degree per second). The joint angular velocity (degree per second) is recorded by wearable sensors (inertial movement units) or optical motion sensors (camera).
Joint movement (degree) | 3 year.
  Joint movement (degree) of subjects is recorded by wearable sensors (inertial movement unit) or optical motion sensors (camera) during flat ground walking and up/down stairs situation.
Body center of mass sway (millimeter) during testing session | 3 year.
  The shift (millimeter)) of light and motion markers on subject's pelvis recorded by wearable sensors (inertial movement unit) or optical motion sensors (camera) and forceplae during flat ground walking and up/down stairs situation.

SECONDARY OUTCOMES:
Activities-Specific Balance Confidence Scale (ABC scale). | 3 year.
  Clinical assessment scales to identify individuals with a fall risk. The minimum and maximum values are 0% and 100%, and whether higher scores mean a better outcome.
Dizziness Handicap Inventory (DHI). | 3 year.
  Clinical assessment scales that quantifies the impact of dizziness on daily life. The minimum and maximum values are 0 and 100, and whether higher scores mean a worse outcome.
Hospital Anxiety and Depression Scale (HADS). | 3 year.
  Clinical assessment scales to measure anxiety and depression in a general medical population of patients. The minimum and maximum values are 0 and 42, and whether higher scores mean a worse outcome.
Dynamic Gait Index (DGI). | 3 year.
  Clinical assessment scales to test the ability of the participant to maintain walking balance while responding to different task demands, through various dynamic conditions. The minimum and maximum values are 0 and 24, and whether higher scores mean a better outcome.
Tinetti Fall Risk Assessment Tool (Tinetti Scale). | 3 year.
  Clinical assessment scales to test the walking and balance ability to valuate the falling risk. The minimum and maximum values are 0 and 28, and whether higher scores mean a better outcome.
Montreal Cognitive Assessment Taiwanese version (MoCA). | 3 year.
  Cognitive-related assessments. The minimum and maximum values are 0 and 30, and whether higher scores mean a better outcome. The minimum and maximum values are 0 and 24, and whether higher scores mean a better outcome.
Trail Making Test. | 3 year.
  Clinical assessment scales which provide information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning. Longer time consumed means worse performance. An average score for TMT-A is 29 seconds and a deficient score is greater than 78 seconds. For TMT-B, an average score is 75 seconds and a deficient score is greater than 273 seconds.
Digit Span Test. | 3 year.
  Clinical assessment scales to test subject's ability to remember a sequence of numbers that appear on the screen, one at a time. The minimum and maximum values are 0 and 21, and whether higher scores mean a better outcome.
Stroop Test. | 3 year.
  Clinical assessment scales for color recognize.The minimum and maximum values are 1% and 100%, and whether the higher percentage rates mean better performance

CONTACTS AND LOCATIONS:
Overall Officials: Chen Po-Yin, Study Chair — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

REFERENCES:
- [Background] Smith PF. Why dizziness is likely to increase the risk of cognitive dysfunction and dementia in elderly adults. N Z Med J. 2020 Sep 25;133(1522):112-127. PMID 32994621
- [Background] Rubenstein LZ. Falls in older people: epidemiology, risk factors and strategies for prevention. Age Ageing. 2006 Sep;35 Suppl 2:ii37-ii41. doi: 10.1093/ageing/afl084. PMID 16926202
- [Background] Brandt T, Daroff RB. The multisensory physiological and pathological vertigo syndromes. Ann Neurol. 1980 Mar;7(3):195-203. doi: 10.1002/ana.410070302. No abstract available. PMID 6999976
- [Background] Aguirre GK, D'Esposito M. Topographical disorientation: a synthesis and taxonomy. Brain. 1999 Sep;122 ( Pt 9):1613-28. doi: 10.1093/brain/122.9.1613. PMID 10468502
- [Background] Stijntjes M, Pasma JH, van Vuuren M, Blauw GJ, Meskers CG, Maier AB. Low cognitive status is associated with a lower ability to maintain standing balance in elderly outpatients. Gerontology. 2015;61(2):124-30. doi: 10.1159/000364916. Epub 2014 Sep 2. PMID 25196019
- [Background] Roberts JC, Cohen HS, Sangi-Haghpeykar H. Vestibular disorders and dual task performance: impairment when walking a straight path. J Vestib Res. 2011;21(3):167-74. doi: 10.3233/VES-2011-0415. PMID 21558642
- [Background] Camicioli R, Oken BS, Sexton G, Kaye JA, Nutt JG. Verbal fluency task affects gait in Parkinson's disease with motor freezing. J Geriatr Psychiatry Neurol. 1998 Winter;11(4):181-5. doi: 10.1177/089198879901100403. PMID 10230996
- [Background] O'Shea S, Morris ME, Iansek R. Dual task interference during gait in people with Parkinson disease: effects of motor versus cognitive secondary tasks. Phys Ther. 2002 Sep;82(9):888-97. PMID 12201803
- [Background] Sheridan PL, Solomont J, Kowall N, Hausdorff JM. Influence of executive function on locomotor function: divided attention increases gait variability in Alzheimer's disease. J Am Geriatr Soc. 2003 Nov;51(11):1633-7. doi: 10.1046/j.1532-5415.2003.51516.x. PMID 14687395
- [Background] Toulotte C, Thevenon A, Fabre C. Effects of training and detraining on the static and dynamic balance in elderly fallers and non-fallers: a pilot study. Disabil Rehabil. 2006 Jan 30;28(2):125-33. doi: 10.1080/09638280500163653. PMID 16393843
- [Background] Holtzer R, Mahoney JR, Izzetoglu M, Izzetoglu K, Onaral B, Verghese J. fNIRS study of walking and walking while talking in young and old individuals. J Gerontol A Biol Sci Med Sci. 2011 Aug;66(8):879-87. doi: 10.1093/gerona/glr068. Epub 2011 May 17. PMID 21593013
- [Background] Chen PY, Wei SH, Hsieh WL, Cheen JR, Chen LK, Kao CL. Lower limb power rehabilitation (LLPR) using interactive video game for improvement of balance function in older people. Arch Gerontol Geriatr. 2012 Nov-Dec;55(3):677-82. doi: 10.1016/j.archger.2012.05.012. Epub 2012 Jul 15. PMID 22795360
- [Background] Borges SM, Radanovic M, Forlenza OV. Correlation between functional mobility and cognitive performance in older adults with cognitive impairment. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2018 Jan;25(1):23-32. doi: 10.1080/13825585.2016.1258035. Epub 2016 Dec 9. PMID 27934540
- [Background] Koh DH, Lee JD, Lee HJ. Relationships among hearing loss, cognition and balance ability in community-dwelling older adults. J Phys Ther Sci. 2015 May;27(5):1539-42. doi: 10.1589/jpts.27.1539. Epub 2015 May 26. PMID 26157259
- [Background] Iwasaki S, Yamamoto Y, Togo F, Kinoshita M, Yoshifuji Y, Fujimoto C, Yamasoba T. Noisy vestibular stimulation improves body balance in bilateral vestibulopathy. Neurology. 2014 Mar 18;82(11):969-75. doi: 10.1212/WNL.0000000000000215. Epub 2014 Feb 14. PMID 24532279
- [Background] Fujimoto C, Yamamoto Y, Kamogashira T, Kinoshita M, Egami N, Uemura Y, Togo F, Yamasoba T, Iwasaki S. Noisy galvanic vestibular stimulation induces a sustained improvement in body balance in elderly adults. Sci Rep. 2016 Nov 21;6:37575. doi: 10.1038/srep37575. PMID 27869225
- [Background] Herdman SJ, Tusa RJ, Blatt P, Suzuki A, Venuto PJ, Roberts D. Computerized dynamic visual acuity test in the assessment of vestibular deficits. Am J Otol. 1998 Nov;19(6):790-6. PMID 9831156
- [Background] Whitney SL, Wrisley DM, Brown KE, Furman JM. Is perception of handicap related to functional performance in persons with vestibular dysfunction? Otol Neurotol. 2004 Mar;25(2):139-43. doi: 10.1097/00129492-200403000-00010. PMID 15021773
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Myers AM, Fletcher PC, Myers AH, Sherk W. Discriminative and evaluative properties of the activities-specific balance confidence (ABC) scale. J Gerontol A Biol Sci Med Sci. 1998 Jul;53(4):M287-94. doi: 10.1093/gerona/53a.4.m287. PMID 18314568
- [Background] Myers AM, Powell LE, Maki BE, Holliday PJ, Brawley LR, Sherk W. Psychological indicators of balance confidence: relationship to actual and perceived abilities. J Gerontol A Biol Sci Med Sci. 1996 Jan;51(1):M37-43. doi: 10.1093/gerona/51a.1.m37. PMID 8548512
- [Background] Tinetti ME, Richman D, Powell L. Falls efficacy as a measure of fear of falling. J Gerontol. 1990 Nov;45(6):P239-43. doi: 10.1093/geronj/45.6.p239. PMID 2229948
- [Background] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Shumway-Cook A, Baldwin M, Polissar NL, Gruber W. Predicting the probability for falls in community-dwelling older adults. Phys Ther. 1997 Aug;77(8):812-9. doi: 10.1093/ptj/77.8.812. PMID 9256869
- [Background] Tinetti ME. Performance-oriented assessment of mobility problems in elderly patients. J Am Geriatr Soc. 1986 Feb;34(2):119-26. doi: 10.1111/j.1532-5415.1986.tb05480.x. No abstract available. PMID 3944402
- [Background] Chen KL, Xu Y, Chu AQ, Ding D, Liang XN, Nasreddine ZS, Dong Q, Hong Z, Zhao QH, Guo QH. Validation of the Chinese Version of Montreal Cognitive Assessment Basic for Screening Mild Cognitive Impairment. J Am Geriatr Soc. 2016 Dec;64(12):e285-e290. doi: 10.1111/jgs.14530. Epub 2016 Nov 7. PMID 27996103
- [Background] Gill-Body KM, Beninato M, Krebs DE. Relationship among balance impairments, functional performance, and disability in people with peripheral vestibular hypofunction. Phys Ther. 2000 Aug;80(8):748-58. PMID 10911413
- [Background] Chen PY, Jheng YC, Wang CC, Huang SE, Yang TH, Hsu PC, Kuo CH, Lin YY, Lai WY, Kao CL. Effect of noisy galvanic vestibular stimulation on dynamic posture sway under visual deprivation in patients with bilateral vestibular hypofunction. Sci Rep. 2021 Feb 19;11(1):4229. doi: 10.1038/s41598-021-83206-z. PMID 33608568